CLINICAL TRIAL: NCT06040437
Title: Be-Prox. An Effectiveness Study of Bullying Intervention in Norwegian Kindergartens.
Acronym: Be-Prox
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: University of Tromso (Other); Bjørnafjorden municipality (Unknown); Narvik municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105246
Record Dates: First submitted 2023-09-02; First posted 2023-09-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Bullying of Child
Keywords: Early Childhood and Educational Care; Norway; Bullying intervention; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Be-Prox intervention (Experimental): Training in the 6 Be-Prox module
  Interventions: Behavioral: Be-Prox
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Be-Prox — Be-Prox is an intervention developed to prevent, uncover and handle negative behavior in kindergartens.
  Arms: Be-Prox intervention

SUMMARY:
With an overall aim to ensure a safe and sound kindergarten environment for all Norwegian children in accordance with the Kindergarten Act §§41-43, the objectives of the current project are:

To evaluate the effectiveness of Be-Prox Norway to prevent and handle negative behavior and bullying among peers in Norwegian kindergartens.

To examine implementation factors that promote and inhibit the effectiveness of Be-Prox Norway in Norwegian kindergartens.

To describe the cost-effectiveness of the Be-Prox Norway intervention in Norwegian kindergartens.

To generate knowledge on how the Be-Prox Norway intervention can be aligned and implemented in Norwegian kindergartens.

DETAILED DESCRIPTION:
January 1st, 2021, new additions to the Kindergarten Act came into force in Norway introducing the right for all children to a safe and sound kindergarten environment. According to this act, Norwegian kindergartens shall systematically work to preventing bullying and social exclusion, including adopting a zero-tolerance for violations such as exclusion, bullying, violence, discrimination, and harassment. While relatively little is known about bullying at this age, a growing body of research suggests that bullying occurs also between kindergarten peers and that experiencing bullying at early age is associated with negative consequences.

Currently there are few evidence-based interventions directly targeting bullying among kindergarten peers. Be-Prox, developed for Swiss kindergartens to prevent, uncover and handle negative behavior and bullying in kindergartens have been translated and adjusted to a Norwegian context in a previous pilot study.

The current project is a close collaboration between two Norwegian municipalities, regional centres for child and youth mental health and welfare, and research and educational institutions.

The project aims to evaluate the effectiveness of the Be-Prox Norway in a cluster randomized controlled trial, including process and implementation evaluation and cost-effectiveness analyses. Hence the project complies with the current call through introducing research on tools, systems and models that promote evidence-based practices in Norwegian kindergartens in general, and to prevent negative acts and bullying between kindergarten peers in particular.

If proven effective, Be-Prox Norway can be offered to kindergartens nationwide as evidence-based practice to prevent, uncover and handle negative behavior and bullying among Norwegian kindergarten peers.

ELIGIBILITY:
Inclusion Criteria:

* Children born 2018-2020 in kindergartens enrolled to the Be-Prox project and with parental consent to participate.
* Personnel i Norwegian kindergartens enrolled in the Be-Prox project and who consent to participate.
* Parents of children in kindergartens enrolled to the Be-prox project

Exclusion Criteria:

* children born 2021-2023
* children with no parental consent to participate

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Total number of negative acts children have been exposed to by peers the last months post intervention. | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, primary outcome will be the total number of negative acts the child has been exposed to overall. The range for the specific negative acts is 0-5, the range for negative acts overall is 0-20.
Total number of negative acts children have exposed peers to the last month post intervention. | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, primary outcome will be the total number of negative acts the child has exposed peers to overall. The range for the specific negative acts is 0-5, the range for negative acts overall is 0-20.

SECONDARY OUTCOMES:
Change in number of children being exposed to negative acts overall "2-3 times a months" or more post intervention | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, the secondary outcome will be a binary outcome on 0) not been exposed to negative acts 2-3 months or more and 1) being exposed to negative acts 2-3 times a month or more.
Change in number of children exposing other children to negative acts overall "2-3 times a month" or more. | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, the secondary outcome will be a binary outcome on 0) not been exposed to negative acts 2-3 months or more and 1) being exposed to negative acts 2-3 times a month or more.
Child prosocial bystander behavior post intervention | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  12 item questionnaire, Alsaker 2004
Change in Authoritative climate, post intervention | The last month post Scorers are asked to use "the 4 weeks" as the time frame for their registration of the negative acts, 1 and 2 years after post intervention
  10 item scale, adjusted from Ertesvåg, 2011
Change in personnel self-efficacy beliefs, post intervention | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  5 item scale, adjusted from Fischer, 2019
Change in personnel understanding of bullying among children in kindergartens | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  8 items questionnaire
Specific negative acts the child has been exposed to the last month | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using the set of questions on specific negative acts; physical, verbal, relational and object-related
Specific negative acts the child has exposed peers to the last month | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using the set of questions on specific negative acts; physical, verbal, relational and object-related
Total number of negative acts children have been exposed to by peers the last | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, primary outcome will be the total number of negative acts the child has been exposed to overall. The range for the specific negative acts is 0-5, the range for negative acts overall is 0-20.
Total number of negative acts children have exposed peers to the last month post | Scorers are asked to use "the last 4 weeks" as the time frame for their registration of the negative acts
  Using a set of questions on physical, verbal, relational and object-related negative acts, primary outcome will be the total number of negative acts the child has exposed peers to overall. The range for the specific negative acts is 0-5, the range for negative acts overall is 0-20.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kvestad, Dr, Principal Investigator — NORCE Norwegian Research Center
Locations (4):
- Norway (4):
  - NORCE Norwegian Research Center, Bergen
  - Narvik municipality, Narvik
  - Bjørnafjorden municipality, Os i Østerdalen
  - University of Tromsø, Tromsø

REFERENCES:
- [Derived] Kvestad I, Adolfsen F, Angeles RC, Brandseth OL, Breivik K, Evertsen JG, Foer IK, Haaland M, Homola BM, Hoseth GE, Jonsson J, Kjerstad E, Kyrrestad H, Martinussen M, Moberg A, Moberg K, Skogstrand A, Solberg LR, Aasheim M. Effectiveness of a Bullying Intervention (Be-Prox) in Norwegian Early Childhood and Education Care Centers: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 24;13:e60626. doi: 10.2196/60626. PMID 39447170

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT06040437/SAP_000.pdf